CLINICAL TRIAL: NCT06495528
Title: Bliss DTx Assessment During Course Care Including Port-A-Catheter Setting
Acronym: EPATPAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Butterfly Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A02483-42
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Pain Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BLISS Arm (Experimental): Port-A-Cath setting under local anesthesia combined with Bliss DTx use
  Interventions: Device: Pain management with BLISS DTx
- GOLD STANDARD Arm (Other): Port-A-Cath setting under local anesthesia combined with site standard of care sedation protocol
  Interventions: Other: Pain Management with site standard of care sedation protocol

INTERVENTIONS:
Device: Pain management with BLISS DTx — Bliss DTx is a Digital Therapeutics (DTx) which uses virtual reality augmented with sound and visual stimuli to reduce pain during Port-A-Cath setting
  Arms: BLISS Arm
Other: Pain Management with site standard of care sedation protocol — Sedation (morphine and/or hypnotics and/or anxiolytics and/or conversational hypnosis) reduces pain during Port-A-Cath setting
  Arms: GOLD STANDARD Arm

SUMMARY:
Setting a Port-a Cath is performed in a surgical room, under ambulatory, by a specialist, under local anesthesia. This Port-a Cath is placed in the upper part of the thorax, under the clavicle, and facilitate the administration of certain anticancer drugs or to inject other treatments throughout the course of care.

Setting a Port-a Cath is painful and stressful. In addition to local anesthesia, patients are often offered a sedation: anxiolytics, hypnotics or inhalation of MEOPA.

Butterfly Therapeutics has developed a Digital Therapeutics (DTx) called Bliss DTx which uses virtual reality augmented by sound and visual stimuli. A first clinical study with Bliss DTx showed that the pain level was not significantly different between "Bliss DTx" arm and "MEOPA" arm when performing osteomedullary biopsy.

This study is based on the hypothesis that Bliss DTx use would :

* Be clinically equivalent to a standard protocol (use of hypnotics and/or anxiolytics and/or MEOPA and/or hypnosis conversational) to manage pain during Port-a Cath setting under local anesthesia
* Reduce anxiety before setting a Port-a Cath
* Provide greater satisfaction with the treatment process from patient point of view
* Have organizational impacts, some of which could be economically valued

DETAILED DESCRIPTION:
An implantable catheter port, also called Port-a Cath, is placed in the upper part of the thorax under the clavicle. Setting is performed in a surgical room, under ambulatory, by a specialist, under local anesthesia. This Port-a Cath is set up to facilitate the administration of certain anticancer drugs or to inject other treatments throughout the course of care.

Setting a Port-a Cath is painful and stressful. In addition to local anesthesia, patients are often offered a sedation: anxiolytics as premedication, hypnotics before or during the Port-a Cath setting, inhalation of MEOPA (equimolar mixture of oxygen and nitrogen protoxide, medicinal anxiolytic and analgesic gas , colorless and slightly odorous, mainly used in a hospital environment).

Virtual reality technology allows a person to be immersed in a virtual environment using a device consisting of headset audio and 3D display system. This is a non-invasive device that has an effect on the anxiety and pain level of patients. Butterfly Therapeutics has developed a Digital Therapeutics (DTx) called Bliss DTx which uses virtual reality augmented by sound and visual stimuli. A first clinical study with Bliss DTx which was released in 2021 showed that the pain level was not significantly different between "Bliss DTx" arm and "MEOPA" arm when performing osteomedullary biopsy.

Bliss DTx is also used in everyday practice by many doctors, surgeons, anesthetists and nurses, who do not observe significant pain difference between Bliss DTx and chemical sedations during the acts, but note interesting differences from an organizational point of view between the different methods.

A new evolution of Bliss DTx offers features that allow to increase winnings throughout the course including installation of a Port-a Cath.

This study is therefore based on the hypothesis that Bliss DTx use would :

* Be clinically equivalent to a standard protocol (use of hypnotics and/or anxiolytics and/or MEOPA and/or hypnosis conversational) to manage pain during Port-a Cath setting under local anesthesia
* Reduce anxiety before setting a Port-a Cath
* Provide greater satisfaction with the treatment process from patient point of view
* Have organizational impacts, some of which could be economically valued, contributing to optimization of the entire course care for patients with Port-a Cath setting

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged ≥ 18 years
* Patient with a cancer diagnosis
* Patient with Port-A-Cath setting under ambulatory
* Patient affiliated to or beneficiary of a social security system
* French speaking patient having signed informed consent

Exclusion Criteria:

* Patient with previous Port-A-Cath setting
* Patient with pain perception disorder
* Patient with contraindication to the use of virtual reality (VR) and screens
* Pregnant woman
* Protected patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-05-12 (Estimated); Study Completion 2025-05-12 (Estimated)

PRIMARY OUTCOMES:
Pain level | 1 day
  Maximum pain level during Port-A-Cath setting will be assessed using Visual Analog Scale : from 0 (no pain) to 10 (intolerable)
Patient anxiety | 1 day
  Patient anxiety before Port-A-Cath setting will be assessed with Hamilton score.
  Score 10 to 13: mild depressive symptoms. Score 14 to 17: mild to moderate depressive symptoms. Score greater than 18: moderate to severe depressive
Patient satisfaction | 1 day
  The overall experience score and patient satisfaction will be assessed using the e-Satis questionnaire in ambulatory surgery (MCO CA) at the end of the treatment course. This a specific french questionnaire without global final score. There are only questions with following rating : poor, weak, medium, good, excellent

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No